CLINICAL TRIAL: NCT04006743
Title: The Effect of Expressed Breast Milk, Swaddling and Facilitated Tucking Methods in Reducing the Pain Caused by Orogastric Tube Insertion in Preterm Infants: A Randomized, Controlled Trial
Brief Title: The Nonpharmacological Methods in Reducing the Pain Caused by Orogastric Tube Insertion in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Vildan Apaydin Cirik, Research Asistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2018-3032
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Pain; Preterm; Premature
Keywords: pain; preterm; premature; orogastric tube; newborn nurse
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Intervention Model Description: This study was randomized controlled trial on the effects of combined and alone use of swaddling, expressed breast milk, and facilitated tucking on preterm infants before, during and after OGT insertion procedure. Preterm infants were randomly allocated before the OGT insertion by a neonatal nurse using a random closed envelope manner to one of the six groups: routine care group, swaddling, expressed breast milk, facilitated tucking, swaddling+expressed breast milk, and facilitated tucking+expressed breast milk group. After obtaining parental written consent, neonatal nurse who apply OGT insertion randomized the infant and learned the allocation group. The nurses could not be blinded to the allocation because of the nature of the intervention. However, nurses were blinded to the study hypotheses. Additionally, the outcome assessment of the videos was blinded.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment of the videos was blinded. PIPP score was measured by two specialist pain doctors who were blinded to the study purpose, and to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- The routine care group (No Intervention): In the routine care group, while a neonatal nurse performed the OGT insertion procedure, physiological measurements of the highest value of heart rate and the lowest value of oxygen saturation were recorded by one researcher (the first author) 1 min before the procedure, during the process and after the process in 1st and 2nd minutes acquired for each infant in the unit with an individual monitor.
- The swaddling group (Experimental): In this group, preterm infants were given swaddling method.
  Interventions: Behavioral: The swaddling group
- The expressed breast milk group (Experimental): In this group, preterm infants were given expressed breast milk method.
  Interventions: Behavioral: The expressed breast milk group
- The facilitated tucking group (Experimental): In this group, preterm infants were given facilitated tucking method.
  Interventions: Behavioral: The facilitated tucking group
- The swaddling and expressed breast milk group (Experimental): In this group, preterm infants were given combined swaddling and expressed breast milk method.
  Interventions: Behavioral: The swaddling and expressed breast milk group
- The facilitated tucking and expressed breast milk group (Experimental): In this group, preterm infants were given combined facilitated tucking and expressed breast milk method.
  Interventions: Behavioral: The facilitated tucking and expressed breast milk group

INTERVENTIONS:
Behavioral: The swaddling group — The newborns were placed in a supine position on a 90 cm2 soft fabric for swaddling procedure. The upper side of the bandage was aligned with the shoulder of the newborn. Newborns' arms were put in a flexion position. The top of the body was completely covered with a bandage. The infant's head can move freely. The swaddling procedure took about one minute. In the study, swaddling process was applied 10 minutes before the painful procedure. The swaddled newborns remained in the swaddling during the procedure and for 5 minutes after the procedure.
  Arms: The swaddling group
Behavioral: The expressed breast milk group — In terms of the reliability of the study results, nothing was orally given to the preterm infant at least 30 minutes before the procedure. As recommended in the studies, 2 ml oral breast milk was given to preterm infants before the procedure. In the study, breast milk was given slowly to the upper part of the tongue of each preterm infant from his/her own mother as a single dose before OGT insertion. As a result, preterm was ensured to take all of 2 ml breast milk by reducing the aspiration risk of breastmilk. The breast milk was given without touching the tip of the injector to the newborn's mouth. The preterm infants were not allowed to suck the tip of the injector.
  Arms: The expressed breast milk group
Behavioral: The facilitated tucking group — Facilitated tucking was given in supine position by holding the arm and legs of the preterm infant to the body by the researcher. In line with the literature, facilitated tucking was initiated 3 minutes before OGT insertion in order for the newborn to feel the fetal position and to cope with the painful procedure. The preterm was kept in fetal position during the procedure and for 5 minutes after the procedure.
  Arms: The facilitated tucking group
Behavioral: The swaddling and expressed breast milk group — Swaddling procedure was conducted by the researcher to the preterm infant 10 minutes before the OGT insertion procedure. 2 ml breast milk was administered by the researcher to preterm using a sterile injector as a single dose for 2 minutes before OGT insertion procedure. The preterm was remained in swaddling during the OGT insertion procedure and for 5 minutes after the process.
  Arms: The swaddling and expressed breast milk group
Behavioral: The facilitated tucking and expressed breast milk group — Facilitated tucking method was applied right after giving 2 ml breast milk by the researcher to the preterm 3 minutes before OGT insertion procedure. Preterm newborn remained in facilitated tucking during the procedure and for 5 minutes after the procedure.
  Arms: The facilitated tucking and expressed breast milk group

SUMMARY:
According to the World Health Organization, preterm birth (from 20 to 37 gestation week) is a significant global health problem, as preterm infants represent an estimated 15 million infants per year worldwide. One of the important problems experienced by the preterm infants, leaving their intrauterine environment earlier than normal, while receiving special treatment and care in Neonatal Intensive Care Unit is the painful procedures. Exposure to pain may change preterm infants' brain structure and organization as well as impair brain development through oxygen desaturation, leading to generation of free radicals that can damage fast-growing tissues. For this reason, preterm infants need to be supported and protected more in pain procedures. Orogastric Tube (OGT) is a feeding method that is used to support the nutrition of preterms that cannot be fed orally and causes OGT insertion pain. Although non-pharmacological methods are effective in reducing the pain caused by OGT insertion in preterms, a limited number of studies have been found. There was no study using combined nonpharmacological methods to reduce OGT insertion pain.To evaluate the efficacy of the use of expressed breast milk, swaddling and facilitated tucking methods alone and combination in reducing the pain caused by OGT insertion in preterms. Randomized controlled trial. Three level III neonatal intensive care units in Turkey. Preterm infants born 32-34 weeks of gestation were randomly assigned to six groups: routine care group (n=33), swaddling group (n=30), facilitated tucking (n=32), expressed breast milk (n=31), swaddling+expressed breast milk group (n=30), and facilitated tucking+expressed breast milk group (n=31). OGT insertion included four phases: baseline (the last 1 min of the 30 min without stimuli), OGT insertion, recovery (1 min after OGT insertion), recovery (2 min after OGT insertion). Four phases of OGT insertion procedures were videotaped. Premature infant pain profile (PIPP) score, heart rate, and oxygen saturation were assessed by two independent evaluators who were blinded to the purpose of the study. Data were analyzed by analysis of variance for the multiple repeated measurements, bonferroni, Generalised Estimating Equation logistic regression. 187 preterm infants completed the protocol.

DETAILED DESCRIPTION:
Orogastric tube feeding is a feeding method used to support the feeding of newborns who cannot be fed orally and OGT insertion causes pain. Ottawa Neonatal Pain Interest Group (2015) and the studies have shown that OGT insertion causes acute pain in newborns. It was stated that OGT insertion causes pain in newborns and non-pharmacological methods were effective in reducing this pain. However, there have been no studies in which non-pharmacological methods (expressed breast milk, swaddling and facilitated tucking methods) are alone and in combination with OGT insertion procedural pain for preterm infants. Therefore, the purpose of this study is to evaluate the efficacy of using expressed breast milk, swaddling and facilitated tucking methods together and alone in reducing the pain caused by OGT insertion process in preterm infants. Based on the above literature review and mechanisms, the investigators hypothesized that: (1) Swaddling, expressed breast milk, and facilitated tucking alone could be more effective than routine care on preterm infant pain before, during, and after OGT insertion procedure. (2) Pain occur less frequently before, during, and after OGT insertion procedure in preterm infants treated with combinations of swaddling, expressed breast milk, and facilitated tucking than in those receiving routine care. (3) Combined intervention of swaddling+expressed breast milk, and facilitated tucking+expressed breast milk could be more effective than any single intervention on preterm infant pain before, during, and after OGT insertion procedure.

Preterm infants were recruited by convenience sampling from level III neonatal intensive care units of three hospitals in Turkey/Antalya from November 2017 to 2018. Preterm infants meeting study criteria (n=219) from 2017 to 2018. Participation was refused by 24 parents who did not want their infants to be videotaped data collection (12), refused anything extra done to their infants (n=10), were not interested (n=2) and 8 infants did not need OGT insertion; thus, 187 infants participated in this study. Preterm infants who did participate did not differ significantly in terms of sex, GA, postnatal age, and body weight. To calculate study power, the investigators first determined that the effect size was 0.51, based on the mean Premature Infant Pain Profile (PIPP) scores, respectively, and the correlation (r=0.385) of PIPP scores between the six groups. Based on this effect size and a significance level of 0.05, the study power (two tailed) with 187 infants was 0.99. Based on the between- and within-group variances of PIPP scores during OGT insertion procedures the effect size was 0.33. Thus, a sample size of 187 preterm infants was sufficient. Preterm infants were randomly allocated before the OGT insertion by a neonatal nurse using a random closed envelope manner to one of the six groups: routine care group, swaddling, expressed breast milk, facilitated tucking, swaddling+expressed breast milk, and facilitated tucking+expressed breast milk group. After obtaining parental written consent, neonatal nurse who apply OGT insertion randomized the infant and learned the allocation group. The nurses could not be blinded to the allocation because of the nature of the intervention. However, the outcome assessment of the videos was blinded. OGT insertion procedure was conducted by the clinical nurse in NICU within the scope of treatment for preterm infants in the case when clinical physician was deemed as necessary. The assigned treatment condition was administered by one researcher. In the routine care group, while a neonatal nurse performed the OGT insertion procedure, physiological measurements of the highest value of heart rate and the lowest value of oxygen saturation were recorded by one researcher 1 min before the procedure, during the process and after the process in 1st and 2nd minutes acquired for each infant in the unit with an individual monitor. In the swaddling group, swaddling process was applied 10 minutes before the painful procedure. The swaddled newborns remained in the swaddling during the procedure and for 5 minutes after the procedure. In the study, breast milk was given slowly to the upper part of the tongue of each preterm infant from his/her own mother as a single dose before OGT insertion. In the expressed breast milk group, preterm was ensured to take all of 2 ml breast milk by reducing the aspiration risk of breastmilk. The breast milk was given without touching the tip of the injector to the newborn's mouth. The preterm infants were not allowed to suck the tip of the injector. In the facilitated tucking group, facilitated tucking was initiated 3 minutes before OGT insertion in order for the newborn to feel the fetal position and to cope with the painful procedure. The preterm was kept in fetal position during the procedure and for 5 minutes after the procedure. In the combined swaddling and expressed breast milk group, swaddling procedure was conducted by the researcher to the preterm infant 10 minutes before the OGT insertion procedure. 2 ml breast milk was administered by the researcher to preterm using a sterile injector as a single dose for 2 minutes before OGT insertion procedure. In the combined facilitated tucking and expressed breast milk group, facilitated tucking method was applied right after giving 2 ml breast milk by the researcher to the preterm 3 minutes before OGT insertion procedure. The Premature Infant Pain Profile (PIPP) scale was used for the pain assessment. Physiological indicators were continuously monitored and behavioral indicators (facial images) were videotaped by a real-time colour video recorder. The digital camera was fixed at a certain angle via the tripod 30 minutes before the procedure. Pain was scored from videotapes of infants' faces 10 min before, 2 min during, and 5 min after OGT insertion procedures. PIPP score was measured by two specialist pain doctors who were blinded to the study purpose, and to the study group allocation. The inter-rater reliability of the Premature Infant Pain Profile ranged from 0.97-0.99 (0.97 for baseline [phase 1], 0.97 phase 2, 0.98 phase 3, 0.99 phase 4, respectively). All preterm infants, heart rate and oxygen saturation were measured using an electrocardiographic bedside monitor and continuously recorded by custom computer software.

Each OGT insertion included four phases: (1) Baseline: 1 min of baseline was collected at the end of the 30 min without stimuli. (2) OGT insertion: conducting the OGT measurement, inserting and fixing OGT (3) Recovery: one min after OGT insertion. (4) Recovery: two min after OGT insertion. Heart rate, oxygen saturation, and PIPP scores were evaluated by four phases.

For the statistical analysis of the data obtained in the study, SPSS (Statistical Package for Social Science) for Windows 22.0 and SAS software, version 9.4 (SAS Institute Inc., Cary, NC, USA) packaged software were used. In the analysis of the measurements such as heart rate and oxygen saturation taken from the same newborns at different times, both graphical methods and repeated measures analysis of variance were used. Paired-sample t-test was applied to the features found to be significant as a result of repeated measures analysis of variance. Advanced analysis of the Bonferroni post-hoc test was also performed. Concordance between the two first evaluators for the PIPP measurements were evaluated using the intraclass correlation coefficient (ICC).

In order to compare the preterm infants with and without pain in six different application groups, those having PIPP values of ≥6 were defined as 1 "pain" and values less than 6 were defined as 0 "no pain". In the analysis of the repeated measure data obtained from the preterm infants in six application groups and at different measurement times, the Generalized Estimating Equation (GEE) method's multiple logistic regression models were used. When the observations are related with each other as in the data with repeated measures, GEE models give more effective and unbiased estimates than ANOVA-based models. Statistical significance was defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* gestational age (GA) between 32 and 34 weeks at delivery
* postnatal age between 3 and 28 days
* being fed with OGT
* not scheduled to receive sedatives, muscle relaxants, or analgesic drugs 24 h before a study session
* having spontaneous breathing
* having breast milk. In this study, GA was defined as the time (in weeks) from the first day of the last menstrual period to date of birth.

Exclusion Criteria:

* history of surgery
* congenital or known genetic anomalies
* disorders affecting brain circulation or cardiovascular system
* severe medical conditions requiring treatment such as sedatives, muscle relaxants, anti-epileptic, or analgesic drugs
* in the condition of fasting
* mother with a history of substance-abuse.

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile (PIPP) | 1 year
  The Premature Infant Pain Profile (PIPP) scale was used for the pain assessment. The primary outcome was the pain score assessed with PIPP scale, a validated and widely used tool to measure procedural pain in preterm infants; It measures pain according to two contextual indicators (gestational age and behavioral state), two physiological indicators (heart rate and oxygen saturation), and three behavioral indicators (brow bulge, eye squeeze, and nasolabial furrow). PIPP scores ≥ 6 are suggested to indicate at least mild pain, and scores ≥ 12 are suggested to indicate moderate-to-severe pain.

SECONDARY OUTCOMES:
Heart Rate | 1 year
  The number of heartbeats per minute was obtained using an electrocardiographic bedside monitor and continuously recorded by custom computer software. An electrocardiographic bedside monitor was inserted into each of the infants.
Oxygen Saturation | 1 year
  Oxygen saturation (SpO2) was obtained using an electrocardiographic bedside monitor and continuously recorded by custom computer software. A separate an electrocardiographic bedside monitor was inserted into each of the infants.
Measurement of incidence of adverse events | 1 year
  The safety of different interventions (swaddling, expressed breast milk, facilitated tucking and combined use of them) was assessed by the incidence of adverse events during the study period. The adverse events included: apnea, aspiration, cyanosis, tachycardia, bradycardia, tachypnea, dyspnea. The adverse events were monitored and recorded by specialist neonatal doctors (a total of three doctors, one from each of three hospitals) who were blind to the purpose of the study. In case of a side effect, it was planned for the specialist neonatal doctor to stop the intervention immediately and to intervene.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date